CLINICAL TRIAL: NCT00278564
Title: High Dose Cyclophosphamide & ATG With Hematopoietic Stem Cell Transplantation in Patients With Refractory Idiopathic Inflammatory Myopathy Diseases: A Phase I Trial
Brief Title: Stem Cell Transplantation in Idiopathic Inflammatory Myopathy Diseases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: high relapse rate
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU FDA IIM.Auto2003
Record Dates: First submitted 2006-01-15; First posted 2006-01-18 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2017-06

CONDITIONS: MYOPATHY
MeSH Terms: conditions — Muscular Diseases | interventions — Hematopoietic Stem Cell Transplantation; Cyclophosphamide; Mesna; thymoglobulin; Methylprednisolone; Granulocyte Colony-Stimulating Factor; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hematopoietic stem cell transplantation (Experimental): Intervention as hematopoietic stem cells transplantation after conditioning regimen: Autologous hematopoietic stem cells will be injected after conditioning regimen
  Interventions: Biological: Hematopoietic stem cell transplantation; Drug: Cyclophosphamide; Drug: Mesna; Drug: ATG(rabbit); Drug: Methylprednisolone; Drug: G-CSF; Drug: Rituxan

INTERVENTIONS:
Biological: Hematopoietic stem cell transplantation — Autologous hematopoietic stem cell transplantation
Drug: Cyclophosphamide
  Other Names: Cytoxan
Drug: Mesna
Drug: ATG(rabbit)
Drug: Methylprednisolone
Drug: G-CSF
Drug: Rituxan

SUMMARY:
Myositis is a disease, believed to be due to immune cells, cells which normally protect the body, but are now attacking the muscles and other organ systems within body. As a result, the affected muscles and organs fail to work properly causing weakness, difficulty swallowing, skin rash, respiratory problems, heart problems, joint stiffness, soft tissue calcification and vasculitis (blood circulation problems). The likelihood of progression of this disease is high. This study is designed to examine whether treating patients with high dose cyclophosphamide (a drug which reduces the function of the immune system) and ATG (a protein that kills the immune cells that are thought to be causing this disease), followed by return of previously collected blood stem cells will stop the progression of myositis.

DETAILED DESCRIPTION:
Conditioning Regimen (In order to assure sterility testing, a minimum of 14 days will be required between stem cell collection and starting the conditioning regimen).

The conditioning regimen is outlined in below:

Cyclophosphamide 50 mg/kg/day will be given IV over 1 hour in 250 cc of normal saline on day -5, -4, -3, and -2. If actual weight is < ideal weight, cyclophosphamide will be given based on actual weight. If actual weight is > ideal weight, cyclophosphamide will be given as adjusted ideal weight. Adjusted ideal weight = ideal weight + 40% (actual weight minus ideal weight).

Mesna 50mg/kg/day will be given IV over 24 hours in 250 cc of normal saline or D5W starting at 10AM each dose. Weight base is calculated same as cyclophosphamide as above.

1ATG (rabbit) 0.5 mg/kg on day -6 and 1mg/kg on day -5, -4, -3, -2 and -1 (total 5.5mg/kg, no dose adjustment) will be given IV over 10 hours in 250 cc of normal saline beginning at least 1 hour after infusion of cyclophosphamide. Premedicate with acetaminophen 650 mg po and diphenhydramine 25 mg po/IV 30 minutes before the infusion.

Methylprednisolone- A suggested dose of 250mg IV should be administered 30 minutes before each ATG infusion.

Hydration- A suggested rate of 125 cc/hr NS should be given starting 6 hours before the first cyclophosphamide dose and continued until 24 hours after the last cyclophosphamide dose. The rate of hydration will be aggressively adjusted. BID weights will be obtained. Amount of fluid can be modified based on patient's fluid status. Minimum target urine output is 2 liters/m2/day

G-CSF 5 mcg/kg/day will be given subcutaneously and continued until the absolute neutrophil counts reaches at least 500/µl.

Rituxan 500 mg will be given IV on the day before the first dose of ATG and the day after stem cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years and ≤ 65 years at the time of pretransplant evaluation.
2. An established diagnosis of polymyositis, dermatomyositis, juvenile polymyositis/dermatomyositis, and myositis associated with other collagen diseases. Diagnosis requires electrophysiological studies and histopathologic features. MRI evidence of muscle inflammation or histological evidence of active myositis is mandatory at entry. If patient had dermatomyositis/polymyositis associated with malignancy, the patient has to be free of malignancy for 5 years and considered to be cured.
3. Patients who failed conventional treatment of at least 3 months duration including high-dose corticosteroids (equivalent dosage of prednisone >1.0 mg/kg/day to start), and must also have failed two or more of the followings: cyclophosphamide, azathioprine, 6-MP, methotrexate, tacrolimus, cyclosporin A, mycophenolate mofetil, TNF inhibitor (e.g. etanercept), IVIG or any other immunosuppressive drugs or immune modulating drugs.
4. Failure is defined by (one or more of the following) (not caused by unrelated conditions):

   * Persistent muscle weakness (grade 4/5 or worse by MRC) with elevation of muscle derived enzymes (CPK, aldolase)
   * Worsening pulmonary function especially %VC or DLCo > 15% over 12 months indicating active alveolitis.
   * Abnormal EKG or echocardiographic evidence of cardiomyopathy.
   * Presence of progressive joint contracture, progressive calcinosis, vasculitis, or skin ulcers in juvenile dermatomyositis/polymyositis.

Exclusion Criteria:

1. Poor performance (PS) status (ECOG >2) at the time of entry, unless decline of PS is due to the disease itself.
2. Significant end organ damage such as (not caused by IIM):

   * LVEF <40% or deterioration of LVEF during exercise test on MUGA or echocardiogram.
   * Untreated life-threatening arrhythmia.
   * Active ischemic heart disease or heart failure.
   * DLCo <40% or FEV1/FEV < 50%.
   * Serum creatinine >2.5 or creatinine clearance <30ml/min.
   * Liver cirrhosis, transaminases >3x of normal limits or bilirubin >2.0 unless due to Gilbert disease.
3. HIV positive.
4. Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive treatment.
5. Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as (but not limited to) head and neck cancer, or stage I or II breast cancer will be considered on an individual basis.
6. Positive pregnancy test, inability or unable to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
7. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
8. Inability to give informed consent.
9. Major hematological abnormalities such as platelet count less than 100,000/ul, ANC less than 1000/ul.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Hematopoietic Stem Cell Transplantation: Intervention as autologous hematopoietic stem cell transplantation after conditioning regimen
  Hematopoietic stem cell transplantation: Autologous hematopoietic stem cell transplantation
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplantation
Started | 7
Completed | 3
Not Completed | 4
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Survival
Time Frame: up to 5 years
Population: All participants who underwent stem cell transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: 6 months, 1 year, then yearly up to 5 years post transplant
Arm/Group | Hematopoietic Stem Cell Transplantation
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=7)
Sinusitis (Infections and infestations) | 2 (2) — Two patients had sinusitis treated with oral antibiotics and IVIG and resolved with treatment.
Viral infection (General disorders) | 1 (2) — one hospitalization for transient nausea, vomiting and diarrhea-- no documented etiology.
hypokalemia (General disorders) | 1 (1) — One patient had transient asymptomatic grade 4 hypokalemia during transplant.

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes